CLINICAL TRIAL: NCT03760575
Title: Pembrolizumab in Combination With Chemotherapy and Image-Guided Surgery for Malignant Pleural Mesothelioma (MPM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 07518; 831466 (Other: UPenn IRB)
Record Dates: First submitted 2018-09-26; First posted 2018-11-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Mesotheliomas Pleural
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — pembrolizumab; Indocyanine Green; Surgery, Computer-Assisted; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab with image-guided surgery and chemotherapy (Experimental)
  Interventions: Drug: Pembrolizumab; Procedure: Indocyanine Green (ICG) Image-Guided Surgery; Drug: Cisplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg via IV infusion every 3 weeks for 2 cycles 3 pre-surgery, for 4 cycles post-surgery and then every 3 weeks during maintenance.
  Other Names: MK-3475
Procedure: Indocyanine Green (ICG) Image-Guided Surgery — Standard surgery with image guided resection.
Drug: Cisplatin — 75 mg/m2 every 3 weeks via IV infusion for 4 cycles post-surgery.
Drug: Pemetrexed — 500 mg/m2 every 3 weeks via IV infusion for 4 cycles post-surgery.

SUMMARY:
The study is a single-arm phase I trial to evaluate the safety, feasibility, and preliminary efficacy of the addition of pembrolizumab and image-guided resection to surgical therapy and chemotherapy for malignant pleural mesothelioma (MPM).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Be 18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment OR Is taking chronic systemic steroids (in doses exceeding 10 mg daily of prednisone equivalent) within 7 days prior to the first dose of trial treatment. (Note: Subjects with asthma or chronic obstructive pulmonary disease that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.)
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to ICG or pembrolizumab or any of their excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known metastatic disease and/or disease that is otherwise determined to be unresectable.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Evidence of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Study related adverse events (AEs) | Each subjects will be assessed for AEs from the time of their first study treatment until 30 days after the end of their treatment for AEs and until 90 days after their last treatment for serious AEs (study treatment may last for up to 1 year)
  Study related adverse events (AEs)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Each subject will be assessed for PFS from the time of their first study treatment until the date when they have documented disease progression or death (whichever comes first), or until the study is completed (estimated 2 years for study completion)
  Progression-free survival (PFS)
Overall survival (OS) | Each subject will be assessed for OS from the time of their first study treatment until the date when they have documented disease progression or death (whichever comes first), or until the study is completed (estimated 2 years for study completion)
  Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Corey Langer, MD, Principal Investigator — University of Pennsylvania Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided